CLINICAL TRIAL: NCT00355732
Title: Chronic Obstructive Pulmonary Disease and Weaning From Mechanical Ventilation in Difficult to Wean Patients; Randomized Prospective Study
Brief Title: Chronic Obstructive Pulmonary Disease and Weaning From Mechanical Ventilation in Difficult to Wean Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Josip Benčević General Hospital (Other)
Collaborators: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2006-07-23; First posted 2006-07-25 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-07

CONDITIONS: Respiratory Failure
Keywords: Respiration; COPD; Mechanical Ventilation; Ventilator Weaning; Respiratory Failure; ICU; Pressure Support Ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration; Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Procedure: Weaning from mechanical ventilation

SUMMARY:
To evaluate and compare two methods of weaning from mechanical ventilation in patients with chronic obstructive pulmonary disease (COPD) where the extubation failed.

DETAILED DESCRIPTION:
A prospective, randomized trial was performed in a multidisciplinary Intensive Care Unit (ICU) for the duration of 2 years. A total of 136 COPD patients who required mechanical ventilation longer than 24 h fulfilled the inclusion criteria and they present the research sample. After fulfilling the criteria for weaning, patients were randomized to a 2-h spontaneous breathing trial with either T-tube or pressure support ventilation (PSV). The patients with successful 2-h trial were extubated and were excluded from further research. Patients with 2-h trial failure were defined as difficult to wean, they had mechanical ventilation reinstated and the same weaning procedure was repeated after 24 h, if the patient again fulfilled the weaning criteria. In these patients, two methods of weaning were compared according to the patients clinical characteristics, objective parameters and procedure outcome.

31 (47%) patient with T-tube and 32 (46%) patients with PSV had 2-h trial failure. Of those patients, successful extubation was in 17 (56%) patients with T-tube and in 23 (72%) with PSV (P <0.001), whereas extubation failure was in 14 (44%) patients with T-tube and in 9 (28%) patients with PSV (P <0.001). Mechanical ventilation duration was 186.7 h with T-tube and 163.2 h with PSV (P <0.001), time spent in ICU was 240.7 h with T-tube and 210.2 h with PSV (P <0.001).

In patients with COPD who failed the 2-h spontaneous breathing trial, based on parameters of procedure outcome, high advantage of PSV method was confirmed.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* exacerbation of dyspnea <2 weeks
* signs of respiratory muscle dysfunction

Exclusion Criteria:

* non COPD patients
* age <18 years
* tracheotomy
* MV duration shorter than 24h
* use of MV on admission to the ICU or transfer to some other ICU for treatment continuation
* patients who died or weaning from MV was discontinued because of another associated disorder
* central nerve system disorders unrelated to hypercapnic encephalopathy or hypoxemia
* cardiac arrest within 5 days
* patients scheduled for organ donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Matić, MD PhD, Study Chair — Department of Anesthesiology and Intensive Care, Dr. Josip Benčević General Hospital, Slavonski Brod, Croatia
Locations (2):
- Croatia (2):
  - Dr. Josip Benčević General Hospital, Slavonski Brod
  - Clinic Hospital Center Zagreb, Zagreb